CLINICAL TRIAL: NCT05584319
Title: EMPAGUM: Effects of Empagliflozin on Gut Microbiota in Heart Failure With a Preserved Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhijun Sun (Other)
Responsible Party: Sponsor-Investigator, Zhijun Sun, Director of the second Department of cardiovascular medicine, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022PS999K
Record Dates: First submitted 2022-10-08; First posted 2022-10-18 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Gut Microbiota; SGLT2 Inhibitor; Myocardial Fibrosis; Short-chain Fatty Acids; Derived Metabolite
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin group (Experimental): Subjects in Empagliflozin group take in 10Mg Empagliflozin per day.
  Interventions: Drug: Empagliflozin 10 Mg
- Blank control group (No Intervention): Subjects in Blank control group will not receive Empagliflozin or other sglt-2 inhibitors.

INTERVENTIONS:
Drug: Empagliflozin 10 Mg — subjects in Empagliflozin group takes Empagliflozin 10mg per day
  Other Names: Empagliflozin
  Arms: Empagliflozin group

SUMMARY:
Empagliflozin was recommended for patients with heart failure with reduced ejection fraction (HFrEF) in 2021 European Society of Cardiology (ESC) guidelines (Class of Recommendation Ia) and patients with heart failure with preserved ejection fraction (HFpEF) in 2022 American Heart Association (AHA) guidelines (Class of Recommendation IIa). However, the physiopathologic mechanisms in its effects on HFpEF are not clear. Studies illustrate that gut microbiota plays an essential role in the progress of the heart failure. Studies on mice found that sodium-glucose cotransporter-2 inhibitors (sglt-2i) could affect the intestinal microbiota in mice. The purpose of this study is to clarify the changes of gut microbiota in the patients with HFpEF taking Empagliflozin and explore the role of gut microbiota in this process.

DETAILED DESCRIPTION:
As one of the most important cardiovascular diseases, heart failure is characterized by high incidence and high fatality rate. Heart failure with reduced ejection fraction (HFrEF) has been widely researched for decades and its clinical treatments have been improved remarkably. However, patients with non-reduced ejection fraction accounts for more than 50% of the whole group, especially patients with HFpEF. As for its complicated mechanism as well as normally less serious symptoms, its clinical treatments were not detailed enough before.

Patients with heart failure often have decreased cardiac output combined with peripheral circulation congestion, leading to intestinal ischemia and edema. In this case, the intestinal barrier function is weakened, the intestinal wall permeability increases, the bacterial flora is displaced, and more harmful metabolites would also enter the blood circulation through the weakened intestinal mucosal barrier, inspiring more inflammatory substances and aggravating the states of heart failure.

Empagliflozin is a sodium-glucose transporter 2 (sglt-2) inhibitor, which can inhibit the reabsorption of glucose in the kidney, discharge excessive glucose from the urine, and reduce blood glucose. It is a new type of hypoglycemic drugs. However, as the study progressed, the effect of sglt-2 inhibitors extends. In fundamental and animal trials, sglt-2 inhibitors were found to reduce sodium uptake, inhibit NO synthesis, improve cardiac energy metabolism, and inhibit cardiac inflammation. In the 2021 ESC heart failure guidelines, sglt-2 inhibitors have been included in the "new quadruple" therapy to target patients with HFrEF. Moreover, in the newly published EMPEROR-preserved study, Empagliflozin still achieved very good efficacy in ejection fraction-preserved heart failure, reducing the composite endpoint event by 21%. The mechanisms by which sglt-2 inhibitors act on heart failure have not been fully resolved, and in basic studies, sglt-2 inhibitors were found to affect the intestinal microbiota in mice.

Based on the emerging importance of intestinal microbiota in the process of heart failure, and the impacts of sglt-2 inhibitors on intestinal microbiota and heart failure. It is necessary to clarify the changes of gut microbiota in the patients with non-reduced ejection fraction taking Empagliflozin and explore the role of gut microbiota in this process.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, BMI 18.5-27.9kg/m.
2. Patients with heart failure and EF>40%, New York Heart Association classification ( NYHA) class II-IV and evidence of structural heart disease (i.e. left ventricular hypertrophy or left atrial enlargement by the recent echocardiogram within the last 12 months before enrollment).
3. NT-proBNP≥300 pg/ml for patients without AF, or ≥600 pg/ml for patients with atrial fibrillation (AF).
4. Signed and dated written informed consent form (ICF)

Exclusion Criteria:

* 1.Current use or prior use of a SGLT-2 inhibitor in 3 months. 2.Patients with type 1 diabetes mellitus. 3.History of ketoacidosis. 4.Impaired renal function with estimated glomerular filtration rate (eGFR)<20ml/min/1.73m².

  5.On a diet or with a recent diet plan adjustment. 6.Have gastrointestinal diseases which in active stages (e.g. malabsorptive conditions such as irritable bowel syndrome, coeliac).

  7.Combination of sever infectious diseases (e.g. Severe myocarditis, severe pneumonia, and severe urinary tract infection ).

  8.Acute decompensated heart failure. 9.Severe diseases in other systems (e.g. severe liver insufficiency, moderate-severe anemia, malignant tumors, hematological diseases).

  10.Known or suspected allergy to the active or inactive ingredients of the drug under study.

  11.Admitted percutaneous coronary intervention (PCI), or cardiac surgery, cardiac resynchronization (CRT), or other surgery within the past 90 days.

  12.Arranging to receive cardiovascular revascularization (percutaneous intervention or surgery) or major heart surgery (coronary artery bypass transplantation, valve replacement, ventricular aids, heart transplantation, CRT or any other surgery requiring thoracotomy or transcatheter aortic valve replacement) in 30 days.

  13.Symptomatic hypotension with systolic pressure ≤ 90mmHg. 14.Systolic pressure ≥ 180mmHg which cannot be controlled with drugs. 15.Currently enrolled in another investigational device or drug trial. 16.Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
intestinal microbiota diversity | 6 months
  the changes of Alpha diversity and Beta diversity of intestinal microbiota in samples

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 6 months
  Mace is defined as cardiovascular death and cardiovascular related readmission
N-terminal prohormone of B-type natriuretic peptide ( NT-proBNP ) | 6 months
  Changes of NT-proBNP in 6 months
soluble suppression of tumorigenicity 2 (sST2） | 6 months
  Changes of sST2 in 6 months
serum SCFAs level | 6 months
  Changes of serum SCFAs level in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: 10027 10027, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No